CLINICAL TRIAL: NCT06624046
Title: Circadian Mechanisms of Glycemic Control and Cardiovascular Risk in Adults With Type 1 Diabetes
Brief Title: Circadian Mechanisms, Glucose, and CV Risks in T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pamela Martyn-Nemeth, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-0886; R01HL174738 (NIH)
Record Dates: First submitted 2024-09-27; First posted 2024-10-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: sleep; cardiovascular disease risk; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single arm, pretest, post-test design using a sleep stability intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Sleep stability intervention
  Interventions: Behavioral: Sleep stability intervention

INTERVENTIONS:
Behavioral: Sleep stability intervention — The sleep stability intervention will consist of three theory-based intervention components our team has developed and used in prior interventions: 1) self-monitoring using a wearable sleep tracker (Fitbit). This is well-liked by participants and increases awareness of their sleep goals. 2) Accountability coaching via weekly check-ins and daily monitoring of participants' wearable sleep tracking data and a coaching protocol.

SUMMARY:
People with type 1 diabetes are disproportionately affected by cardiovascular disease (CVD). Short and irregular sleep have been associated with cardiovascular risk in this population. Improving sleep regularity has been associated with improved glycemic markers however mechanisms by which improving sleep regularity improves metabolic and cardiovascular health is not known. The investigators propose to conduct a mechanistic study using a sleep stability manipulation. This proposal will advance the understanding of mechanisms by which improving sleep regularity influences glycemic control and cardiovascular risk in T1D.

DETAILED DESCRIPTION:
People with type 1 diabetes (T1D) are disproportionately affected by cardiovascular disease (CVD). CVD is a leading cause of death in T1D, contributing to 40% of mortality. Sleep is recognized by both the American Heart Association and the American Diabetes Association as a critical health behavior to maintain glycemic control and reduce CVD risk. Short and/or irregular sleep have been associated with reduced glycemic control and non-dipping blood pressure in T1D, both of which are predictors of CV events. Emerging data suggest that behavioral sleep interventions targeting short or irregular sleep led to improved glycemic parameters. However, little is known about the mechanism by which improving sleep duration and/or regularity improves glycemic control and reduces CV risk in T1D. The investigators and others have shown that people with T1D often experience poor sleep health, including inadequate sleep duration, sleep irregularity, and poor sleep quality. The goals of this study are to examine the mechanisms by which improving sleep regularity through behavioral sleep intervention affects glycemic control and CVD risks in T1D adults. The investigators propose to extend our previous research by conducting a mechanistic study using a sleep stability manipulation. The investigators hypothesize that sleep stability impacts glycemic control and CV outcomes by improving circadian regulation. The investigators will conduct a 4-week behavioral sleep stability intervention in 100 T1D adults with irregular sleep, utilizing a sleep pre/post design. Circadian regulation will be assessed by dim-light melatonin onset (DLMO), melatonin metabolite amplitude (overnight urinary 6-sulfatoxymelatonin levels), actigraphy-derived rest-activity rhythm, endothelial cell CLOCK gene mRNA expression, and known zeitgebers of the central and peripheral circadian clocks (light exposure, meal timing). Main glycemic outcomes will be assessed by CGM, A1C, and assessment of insulin sensitivity. Main CV outcomes will include 24h blood pressure and endothelial FMD and other secondary vascular measures (pulse wave velocity, carotid intima media thickness, and echocardiographic parameters). Sleep will be objectively recorded. All parameters will be measured at baseline and end of intervention. This proposal will advance the understanding of mechanisms by which improving sleep regularity influences glycemic control and cardiovascular risk in T1D.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-50 years with a clinical diagnosis of T1D for at least one year
* Report habitual sleep irregularity ≥1 hour/week
* Desire to improve sleep, and own a smartphone (Android or iPhone)

Exclusion Criteria:

* Self-reported A1C within the past 6 months ≥10%
* insomnia symptoms defined as Insomnia Severity Index score ≥15
* history of restless leg syndrome
* history of severe hypoglycemia (defined as hypoglycemic episode that results in loss of consciousness, seizure, or requiring emergency room visit or hospitalization) within the past 6 months
* rotating shift or night work or routinely sleeping after 3 AM.
* use of sleep medications/aids, significant medical comorbidities (such as heart failure, cirrhosis, chronic obstructive pulmonary disease requiring oxygen, active treatment for cancer, on renal replacement therapy [dialysis])
* depression (Patient Health Questionnaire 8 [PHQ-8] score ≥15)
* history of stroke with neurological deficits
* pregnant, breast feeding, or planning pregnancy, as sleep and glucose are known to change during pregnancy and breastfeeding.
* Allergy to lidocaine Participants who passed the first screen by phone will be scheduled for a consenting visit at UIC

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic status | From enrollment to week 12
  Continuous glucose monitor (CGM)
Glycemic control | From enrollment to week 12
  Hemoglobin A1C
Insulin sensitivity | From enrollment to week 12
  Insulin sensitivity

SECONDARY OUTCOMES:
Circadian regulation DLMO | enrollment to week 12
  dim-light melatonin onset (DLMO)
Circadian regulation Melatonin | Enrollment to week 12
  Melatonin metabolite amplitude
Circadian regulation actigraphy | enrollment to week 12
  actigraphy-derived rest activity rhythm
Circadian regulation CLOCK gene | enrollment to week 12
  endothelial cell CLOCK gene mRNA expression
Circadian regulation light | enrollment to week 12
  light exposure
Circadian regulation meals | enrollment to week 12
  Meal timing
Cardiovascular outcome blood pressure | enrollment to week 12
  24 hour blood pressure
Cardiovascular outcome endothelial function | enrollment to week 12
  endothelial flow-mediated dilation
Cardiovascular outcome arterial stiffness | enrollment to week 12
  pulse wave velocity
Cardiovascular outcome echocardiogram | enrollment to week 12
  echocardiogram
Cardiovascular outcome CIMT | enrollment to week 12
  carotid intima lining thickness (CIMT)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
The plans for data sharing are currently under review.